CLINICAL TRIAL: NCT05310071
Title: A Phase 3b/4 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Verify the Clinical Benefit of Aducanumab (BIIB037) in Participants With Alzheimer's Disease
Brief Title: A Study to Verify the Clinical Benefit of Aducanumab in Participants With Early Alzheimer's Disease
Acronym: ENVISION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 221AD305; 2022-001671-14 (EudraCT Number)
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — aducanumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aducanumab (Experimental): Participants will receive aducanumab, up to 10 milligrams per kilogram (mg/kg), monthly (once every four weeks), administered as intravenous (IV) infusion.
  Interventions: Drug: Aducanumab
- Placebo (Placebo Comparator): Participants will receive placebo, monthly (once every four weeks), administered as IV infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aducanumab — Administered as specified in the treatment arm.
  Other Names: BIIB037; Aducanumab-avwa; Aduhelm
  Arms: Aducanumab
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to verify the clinical benefit of monthly doses of aducanumab in slowing cognitive and functional impairment as measured by changes in the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) score as compared with placebo in participants with early Alzheimer's disease.

ELIGIBILITY:
Key Inclusion Criteria:

* The participant must have confirmed amyloid beta pathology by cerebrospinal fluid (CSF) or amyloid PET
* Must have a history of subjective memory decline with gradual onset and slow progression over the 6 months before Screening, confirmed by study partner
* The participant must have 1 informant/care partner who, in the Investigator's opinion, has frequent and sufficient contact with the participant (at least 10 hours/week in person or by phone) as to be able to provide accurate information about the participant's cognitive and functional abilities over time
* Must meet all of the following clinical criteria for MCI due to Alzheimer's disease or mild Alzheimer's disease according to National Institute on Aging and Alzheimer's Association (NIA-AA) criteria

  1. Have an MMSE score between 22 and 30 inclusive
  2. Have a CDR memory score >0.5
  3. Have a Clinical Dementia Rating Scale Global Score (CDR-GS) of 0.5 or 1.0
  4. Have a Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) score of 85 or lower indicative of objective cognitive impairment
* Apart from a clinical diagnosis of early Alzheimer's disease, the participant must be in good health as determined by the Investigator based on medical history and screening assessments
* Must consent to apolipoprotein E (ApoE) genotyping. (Note: Participants are not required to be ApoE ε4 carriers)

Key Exclusion Criteria:

* Any uncontrolled medical or neurological/neurodegenerative condition (other than Alzheimer's disease) that, in the opinion of the Investigator, might be a contributing cause of the participant's cognitive impairment
* Clinically significant and/or unstable psychiatric illness within 6 months prior to Screening
* Transient ischemic attack or stroke or any unexplained loss of consciousness within 1 year prior to Screening
* History of severe allergic or anaphylactic reactions or of hypersensitivity to any of the inactive ingredients in the drug product
* Participation in any study with purported disease-modifying effect in Alzheimer's disease within 12 months prior to Screening unless documentation of receipt of placebo is available
* Current use or previous use of medications with a purported disease-modifying effect in Alzheimer's disease, outside of investigational studies
* Use of any medications that, in the opinion of the Investigator, may contribute to cognitive impairment, put the participant at higher risk for AEs, or impair the participant's ability to perform cognitive testing or complete study procedures
* Use of any investigational drug
* Prior exposure to aducanumab either commercially or by participation in a previous study with aducanumab. (Participants are eligible if they did not receive active aducanumab.)
* A negative PET scan result with any amyloid-targeting ligand within 12 months prior to Screening

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1027 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (265):
- United States (130):
  - Gilbert Neurology Partners, PLLC, Gilbert, Arizona
  - Xenoscience Inc., Phoenix, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - HonorHealth Neurology, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Banner Alzheimer's Institute, Tucson, Arizona
  - Health Initiatives Research, Fayetteville, Arkansas
  - Sun Valley Behaivoral Med Center, El Centro, California
  - Neuropain Medical Center, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Irvine Center for Clinical Research, Inc., Irvine, California
  - Mary S. Easton Center for Alzheimer's Disease Research, UCLA, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Anderson Clinical Research, Redlands, California
  - Sutter Health-San Francisco, San Francisco, California
  - University of California San Francisco (PARENT), San Francisco, California
  - The Neuron Clinic, San Marcos, California
  - Syrentis Clinical Research, Santa Ana, California
  - California Neuroscience Research, LLC, Sherman Oaks, California
  - Viking Clinical Research Center, Temecula, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Mountain Neurological Research Center, Basalt, Colorado
  - Yale University, Fairfield, Connecticut
  - Institute for Neurodegenerative Disorders (IND), New Haven, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Howard University Health Sciences, Washington D.C., District of Columbia
  - Neurology of Central Florida Research Center, LLC, Altamonte Springs, Florida
  - JEM Research Institute, Atlantis, Florida
  - Neurology Offices of South Florida, PLLC, Boca Raton, Florida
  - ECommunity Research, LLC, Boca Raton, Florida
  - Nova Clinical Research, LLC, Bradenton, Florida
  - JY Research Institute, Cutler Bay, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Charter Research, LLC, Lady Lake, Florida
  - ARS - Lake Oconee, Lakeland, Florida
  - Medical Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - K2 Medical Research, LLC, Ocoee, Florida
  - K2 Medical Research, LLC, Orlando, Florida
  - K2 Medical Research, Orlando, Florida
  - Headlands Research LLC, Orlando, Florida
  - Conquest Research, Orlando, Florida
  - Quantum Laboratories Inc., Pompano Beach, Florida
  - United Medical Research, Port Orange, Florida
  - Brain Matters Research, Stuart, Florida
  - K2 Medical Research Tampa, Tampa, Florida
  - USF Health Byrd Institute, Tampa, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Great Lakes Clinical Trials, LLC Ravenswood dba Flourish Research, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Alexian Brothers Medical Center - Neuroscience Research Institute, Elk Grove Village, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Fairway, Kansas
  - Ascension Via Christi Research, a division of Ascension Via Christi Hospitals Wichita, Inc., Wichita, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Ochsner Health System PARENT, New Orleans, Louisiana
  - LSU Health Sciences Center Shreveport, Shreveport, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Brigham and Women's Hospital Department of Neurology, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Donald S. Marks, M.D., P.C., Plymouth, Massachusetts
  - Wayne State University - Detroit Medical Center, Detroit, Michigan
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - Center for Memory and Aging, Saint Paul, Minnesota
  - Hattiesburg Clinic, PA, Hattiesburg, Mississippi
  - Sharlin Health and Neurology, Ozark, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - The Cognitive Research Center of New Jersey, Springfield, New Jersey
  - CenExel Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Neurological Associates of Albany, PC, Albany, New York
  - Dent Neurologic Institute, Amherst, New York
  - Social Psychiatry Research Institute (SPRI), Brooklyn, New York
  - New York University Medical Center PRIME, New York, New York
  - Mount Sinai, New York, New York
  - South Shore Neurologic Associates, P.C., Patchogue, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - University of Rochester - PARENT, Rochester, New York
  - Richmond Behavioral Associates ERG Clinical Research - New York PLLC, Staten Island, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - IMA Evaluations LLC, Tarrytown, New York
  - Duke University, Durham, North Carolina
  - AMC Research, LLC, Matthews, North Carolina
  - Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Central States Research, LLC, Tulsa, Oklahoma
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Abington Neurological Associates, LTD, Abington, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Penn Memory Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, East Providence, Rhode Island
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Coastal Neurology PA, Port Royal, South Carolina
  - Neurology Clinic, PC, Cordova, Tennessee
  - Genesis Neuroscience Clinic, Knoxville, Tennessee
  - Senior Adult Specialty Research, Austin, Texas
  - Headlands Research - Brownsville, Brownsville, Texas
  - Kerwin Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Baylor College Of Medicine, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Clinical Trial Network LLC, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - The Memory Clinic, Bennington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Glennan Center for Geriatrics and Gerontology, Norfolk, Virginia
  - National Clinical Research Inc. - Richmond, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Kingfisher Cooperative, LLC, Spokane, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Australia (8):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - KaRa Institute of Neurological Diseases, Macquarie Park, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- Belgium (4):
  - UZ Leuven, Leuven, Flemish Brabant
  - AZ Sint-Jan, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - AZ Groeninge, Kortrijk
- Brazil (5):
  - Trial Tech Tecnologia em Pesquisas com Medicamentos Ltda, Curitiba, Paraná
  - Instituto de Neurologia de Curitiba - Hospital Ecoville, Curitiba, Paraná
  - IMV Pesquisa Neurologica Sociedade Simples Ltda, Porto Alegre, Rio Grande do Sul
  - Instituto do Cerebro do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - IPq-HCFMUSP - Instituto de Psiquiatria do Hospital das Clínicas da FMUSP, São Paulo, São Paulo
- Canada (14):
  - University of Calgary - Heritage Medical Research Clinic, Calgary, Alberta
  - UBC Hospital, Vancouver, British Columbia
  - Centricity Research Halifax, Halifax, Nova Scotia
  - Recherches Neuro-Hippocampe Inc., d/b/a Ottawa Memory Clinic, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program (Neurology Research Inc.), Toronto, Ontario
  - Centricity Research Toronto LMC, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Baycrest Centre for Geriatric Care, Toronto, Ontario
  - Clinique de la Memoire de l'Outaouais, Gatineau, Quebec
  - MoCA Research and Innovation Inc, Greenfield Park, Quebec
  - Montreal Neurological Institute Clinical Research Unit, Montreal, Quebec
  - CHU de Quebec- Hopital de l Enfant Jesus, Québec
- Finland (2):
  - Terveystalo Ruoholahti, Helsinki
  - CRST, Clinical Research Services Turku, Turku
- France (12):
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg, Bas Rhin
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux, Gironde
  - Hôpital La Grave, Toulouse, Haute Garonne
  - Hopital Gui de Chauliac, Montpellier, Herault
  - CHU Rennes - Pontchaillou, Rennes, Ille Et Vilaine
  - CHU Nantes - Hopital Nord Laënnec, Saint-Herblain, Loire Atlantique
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Hôpital Lariboisière, Paris, Paris
  - Hôpital des Chapennes, Villeurbanne, Rhone
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hôpital Broca, Paris
- Germany (18):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - ISPG - Institut fuer Studien zur Psychischen Gesundheit, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Klinikum Bayreuth GmbH- Hohe Warte, Bayreuth, Bavaria
  - Institut fuer Schlaganfall- und Demenzforschung (ISD), Munich, Bavaria
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Zentrum für klinische Forschung Dr.med. Irma Schöll, Bad Homburg, Hesse
  - Universitaetsklinikum Frankfurt Goethe-Universitaet, Frankfurt am Main, Hesse
  - Universitaetsmedizin Goettingen, Göttingen, Lower Saxony
  - Universitaetsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Katholisches Klinikum Bochum gGmbH, Bochum, North Rhine-Westphalia
  - Deutsches Zentrum fuer Neurodegenerative Erkrankungen (DZNE), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Universitaetsklinikum Magdeburg, Magdeburg, Saxony-Anhalt
  - NEUROZENTRUM tempelhof.berlin, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
- Italy (12):
  - Azienda Ospedaliera Card. G. Panico, Tricase, Lecce
  - ASST di Monza, Monza, Milano
  - Fondazione Istituto G.Giglio di Cefalù, Cefalù, Palermo
  - Ospedale di Arzignano, Arzignano VI, Vicenza
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - Azienda Ospedaliera e Universitaria di Perugia, Perugia
  - Fondazione Santa Lucia IRCCS, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno
- Japan (19):
  - National Center For Geriatrics And Gerontology, Obu-shi, Aichi-ken
  - Hakuyokai Kashiwado Hospital, Chiba, Chiba
  - Inage Neurology and Memory Clinic, Chiba, Chiba
  - Southern Tohoku Medical Clinic, Koriyama-shi, Fukushima
  - NHO Hiroshima-Nishi Medical Center, Otake-shi, Hiroshima
  - Himeji Central Hospital Clinic, Himeji-shi, Hyōgo
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Tokushukai Shonan Atsugi Hospital, Atsugi-shi, Kanagawa
  - Tokushukai Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa
  - Teikyo University Hospital, Mizonokuchi, Kawasaki-shi, Kanagawa
  - Rakuwakai Otowa Rehabilitation Hospital, Kyoto, Kyoto
  - NHO Utano National Hospital, Kyoto, Kyoto
  - Katayama Medical Clinic, Kurashiki-shi, Okayama-ken
  - Tokushukai Kishiwada Tokushukai Hospital, Kishiwada-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Midorikai Takesato Hospital, Kasukabe-shi, Saitama
  - Memory Clinic Ochanomizu, Bunkyō City, Tokyo-To
  - National Center of Neurology and Psychiatry, Kodaira-shi, Tokyo-To
  - Tokushukai Yamagata Tokushukai Hospital, Yamagata, Yamagata
- Mexico (5):
  - Hospital Mexico Americano SC, Guadalara, Jalisco
  - Health Pharma Professional Research S.A. de C.V., Mexico City, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Centro de Estudios Clinicos y Especialidades Medicas, S.C., Monterrey, Nuevo León
  - AVIX Investigación Clínica S.C, Monterrey, Nuevo León
- Poland (8):
  - PROMENTE Sp. z o.o., Bydgoszcz, Kujawsko-Pomorskie Województwo
  - Centrum Medyczne NeuroProtect, Warsaw, Mazowieckie Województwo
  - Podlaskie Centrum Psychogeriatrii, Bialystok, Podkarpackie Wojewódctwo
  - Centrum Medyczne Senior, Sopot, Pomorskie Województwo
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie Kliniczny Oddział Neurologii Oddział Udarowy, Lublin
  - NZOZ Wroclawskie Centrum Alzheimerowskie, Wroclaw
  - Nzoz Novo-Med, Katowice, Śląskie Województwo
  - Neuro-Care Gabriela Klodowska, Siemianowice Śląskie, Śląskie Województwo
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (11):
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - Policlinica Gipuzkoa, Donostia / San Sebastian, Guipuzcoa
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Fundacio ACE, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Santa Maria, Lleida
  - Clinica Universidad de Navarra (MAD), Madrid
  - Hospital Victoria Eugenia, Seville
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (3):
  - Skane University Hospital, Malmo, Skåne County
  - Sahlgrenska Universitetssjukhuset, Mölndal Sjukhus, Mölndal, Västra Götaland County
  - Karolinska Universitetssjukhuset, Stockholm
- United Kingdom (11):
  - The University of Edinburgh, Edinburgh, East Lothian
  - Institute of Psychiatry, Psychology and Neuroscience, London, Greater London
  - Re:Cognition Health Ltd (London), London, Greater London
  - Charing Cross Hospital, London, Greater London
  - Park House, Manchester, Greater Manchester
  - Southampton General Hospital, Southampton, Hampshire
  - Moorgreen Hospital, Southampton, Hampshire
  - Brain Health Scotland Life Sciences, Edinburgh, Lothian Region
  - The RICE Centre, Bath, Somerset
  - Glasgow Memory Clinic Ltd, Motherwell, Strathclyde
  - Re Cognition Health Bristol, Bristol

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at the investigative sites in Australia, Belgium, Brazil, Canada, Finland, France, Germany, Italy, Japan, Mexico, Poland, South Korea, Spain, Sweden, United Kingdom, and United States from 02 Jun 2022 to 12 Aug 2024.
Pre-assignment Details: A total of 1027 participants with Alzheimer's Disease (AD) were enrolled and randomized in this study. Of these, 1024 participants were dosed to receive placebo or aducanumab. None of the participants completed the study due to early termination of the study.
Groups:
- Placebo: Participants received placebo, once every four weeks (Q4W), administered as an intravenous (IV) infusion.
- Aducanumab: Participants received aducanumab, up to 10 milligrams per kilogram (mg/kg) of body weight, Q4W, administered as an IV infusion.
Period: Overall Study
Arm/Group | Placebo | Aducanumab
Started (One participant in the placebo arm received drug. This participant was considered in Aducanumab group for safety analysis.) | 344 | 680
Completed | 0 | 0
Not Completed | 344 | 680
Not completed — Death | 0 | 3
Not completed — Adverse Event | 4 | 31
Not completed — Lack of Efficacy - Based on Participant Perception | 0 | 2
Not completed — Protocol Deviation | 2 | 0
Not completed — Randomized by Mistake | 0 | 1
Not completed — Failure to Meet Continuation Criteria | 2 | 0
Not completed — Failure to Meet Randomization Criteria | 1 | 2
Not completed — Site Terminated by Sponsor | 0 | 2
Not completed — Study Terminated by Sponsor | 282 | 559
Not completed — Withdrawal by Participant - Study Visit Burden/Scheduling Conflicts | 14 | 17
Not completed — Withdrawal by Participant - Concern About Study Procedures/Perceived Risks | 2 | 6
Not completed — Withdrawal by Participant Relocation (Moving or Has Moved) | 1 | 3
Not completed — Withdrawal by Participant - Desire for Change in Treatment (Unrelated to Safety/Efficacy) | 8 | 17
Not completed — Withdrawal by Participant - Other | 25 | 30
Not completed — Lost to Follow-up | 2 | 4
Not completed — Reason Not Specified | 1 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who had received at least 1 dose of study treatment (aducanumab or placebo).
Groups:
- Placebo: Participants received placebo, Q4W, administered as an IV infusion.
- Aducanumab: Participants received aducanumab, up to 10 mg/kg of body weight, Q4W, administered as an IV infusion.
- Total: Total of all reporting groups
Arm/Group | Placebo | Aducanumab | Total
Number analyzed (Participants) | 344 | 680 | 1024
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (6.18) | 72.2 (5.81) | 72.3 (5.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 353 | 540
  Male | 157 | 327 | 484
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 39 | 73 | 112
  Race: Black or African American | 3 | 9 | 12
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Race: White | 273 | 533 | 806
  Race: Not Reported Due to Confidentiality Regulations | 26 | 57 | 83
  Race: Other | 0 | 3 | 3
  Race: Multiple: American Indian or Alaska Native and White | 0 | 1 | 1
  Race: Unknown | 1 | 4 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 27 | 51 | 78
  Ethnicity: Not Hispanic or Latino | 293 | 585 | 878
  Ethnicity: Not Reported Due to Confidentiality Regulations | 24 | 43 | 67
  Ethnicity: Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) Score at Week 78
Description: The Clinical Dementia Rate Scale integrates assessments from 3 domains of cognition (memory, orientation, judgment/problem-solving) and 3 domains of function (community affairs, home/hobbies, personal care). Following the caregiver interview and systematic participant examination, the rater assigns a score describing the participant's current performance level in each of these domains of life functioning. The "Sum of boxes" scoring methodology sums the score for each of the 6 domains and provides a value ranging from 0 to 18. Higher scores indicate greater impairment. A positive change from baseline indicates greater impairment.
Time Frame: Baseline, Week 78
Population: FAS included all randomized participants who had received at least 1 dose of study treatment (aducanumab or placebo). Here, 'overall number of participants analyzed' signifies the number of participants available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Participants received placebo, Q4W, administered as IV infusion.
- Aducanumab: Participants received aducanumab, up to 10 mg/kg of body weight, Q4W, administered as IV infusion.
Arm/Group | Placebo | Aducanumab
Number analyzed (Participants) | 6 | 8
score on a scale | 0.67 (0.408) | 1.56 (1.635)

2. Secondary Outcome: Change From Baseline in Integrated Alzheimer's Disease Rating Scale (iADRS) Score at Weeks 78 and 106
Description: The iADRS composite captures a decline in both cognition and daily function. It is a simple linear combination of the Alzheimer's disease assessment scale, cognitive subscale (ADAS-Cog13), and the Alzheimer's disease cooperative study scale for activities of daily living in mild cognitive impairment (ADCS-ADL-MCI). The ADAS-Cog13 scale ranges from 0 to 85 (higher scores indicate worse performance) and the ADCS-ADL-MCI scale ranges from 0 to 53 (higher scores indicate greater independent, healthy functioning). The total score for iADRS scale ranges from 0 to 138, where higher scores indicate better performance.
Time Frame: Baseline, Weeks 78 and 106
Population: FAS included all randomized participants who had received at least 1 dose of study treatment (aducanumab or placebo). Here, 'overall number of participants analyzed' signifies the number of participants available for outcome measure analysis. Assessment was also planned for Week 106 for this outcome measure, but no assessments were conducted at Week 106 due to early termination.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Aducanumab
Number analyzed (Participants) | 3 | 5
score on a scale | -14.667 (4.4869) | -7.796 (6.7805)

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study for Activities of Daily Living in Mild Cognitive Impairment (ADCS-ADL-MCI) Scale Score at Weeks 78 and 106
Description: The ADCS-ADL-MCI scale consists of 17 instrumental items (e.g., shopping, preparing meals, using household appliances, etc) and 1 basic item (getting dressed). Ratings reflect caregiver observations about the participant's actual functioning over the previous month and provide an assessment of change in the functional state of the participant over time. The total score ranges from 0 to 53. Higher scores indicate greater independent, healthy functioning. A positive change from baseline indicates healthy functioning while a negative change from baseline indicates a decline in independent functioning.
Time Frame: Baseline, Weeks 78 and 106
Population: FAS included all randomized participants who had received at least 1 dose of study treatment (aducanumab or placebo). Here 'overall number of participants analyzed' signifies the number of participants available for outcome measure analysis. Assessment was also planned for Week 106 for this outcome measure, but no assessments were conducted at Week 106 due to early termination.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Aducanumab
Number analyzed (Participants) | 3 | 5
score on a scale | -5.0 (3.61) | -0.4 (7.60)

4. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale, Cognitive Subscale (ADAS-Cog13) at Weeks 78 and 106
Description: ADAS-Cog13 comprises both cognitive tasks and clinical ratings of cognitive performance. The cognitive subscale items capture word recall, ability to follow commands, the ability to correctly copy or draw an image, naming, the ability to interact with everyday objects, orientation, word recognition, memory, comprehension of spoken language, word-finding, and language ability, with a measure for delayed word recall and concentration/distractibility. The total score ranges from 0 to 85. Higher scores indicate worse performance. A positive change from baseline indicates decline in cognitive performance.
Time Frame: Baseline, Weeks 78 and 106
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Aducanumab
Number analyzed (Participants) | 3 | 5
score on a scale | 9.667 (0.8844) | 7.396 (2.3262)

5. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) Scale Score at Weeks 78 and 106
Description: The MMSE scale is a performance-based test of global cognitive status. It consists of 11 tasks that assess orientation, word recall, attention and calculation, language abilities, and visuospatial functions. The scores from the 11 tests are combined to obtain the total score, which ranges from 0 to 30. Higher scores indicate better performance. A negative change from baseline indicates decline in cognitive performance.
Time Frame: Baseline, Weeks 78 and 106
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Aducanumab
Number analyzed (Participants) | 3 | 5
score on a scale | -6.0 (1.00) | -1.2 (1.48)

6. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory-10 (NPI-10) Score at Weeks 78 and 106
Description: The NPI-10 is a questionnaire administered to the informant, designed to obtain information on the presence of neuropsychiatric symptoms and behaviors in a participant with Alzheimer's disease. Ten areas are assessed: delusions, hallucinations, agitation/aggression, depression, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability and aberrant motor behavior. The NPI total score ranges from 0 to 120. Higher scores indicate greater impairment. A negative change from baseline indicates improvement (symptom reduction).
Time Frame: Baseline, Weeks 78 and 106
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Aducanumab
Number analyzed (Participants) | 3 | 5
score on a scale | -8.3 (16.20) | -1.8 (6.94)

7. Secondary Outcome: Change From Baseline in Amyloid Positron Emission Tomography (PET) Signal at Weeks 78 and 104
Description: Amyloid PET scan assesses cerebral amyloid load using radiotracers which is standardized into centiloids. Centiloid values on centiloid scale is based on mean composite standardized uptake value ratio (SUVR).
Time Frame: Baseline, Weeks 78 and 104
Population: FAS included all randomized participants who had received at least 1 dose of study treatment (aducanumab or placebo). Here, 'overall number of participants analyzed' signifies the number of participants available for outcome measure analysis. Due to the decision of early termination, only one participant had an amyloid scan at week 78 and data was reported below. In addition, the assessment planned for Week 104 was not performed due to early termination.
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Placebo | Aducanumab
Number analyzed (Participants) | 0 | 1
SUVR |  | -2.360 (NA) — Since there is only 1 participant analyzed, SD was not estimable.

8. Secondary Outcome: Change From Baseline in Tau PET Signal at Weeks 78 and 104
Description: The cerebral tau level was measured by tau PET imaging. Tau PET imaging was conducted using radiotracer. SUVR is a ratio of PET uptake measured in brain region of interest and a disease-free reference region. A higher SUVR is an indication of increased PET radiotracer uptake and worsening disease.
Time Frame: Baseline, Weeks 78 and 104
Population: FAS included all randomized participants who had received at least 1 dose of study treatment (aducanumab or placebo). Here, 'overall number of participants analyzed' signifies the number of participants available for outcome measure analysis. Due to decision of early termination, the Tau PET scan was not performed in any participant at scheduled visits of Weeks 78 and 104.
Arm/Group | Placebo | Aducanumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in CDR-SB Score at Week 106
Description: The CDR integrates assessments from 3 domains of cognition (memory, orientation, judgment/problem-solving) and 3 domains of function (community affairs, home/hobbies, personal care). Following caregiver interview and systematic participant examination, the rater assigns a score describing the participant's current performance level in each of these domains of life functioning. The CDR-SB sums the score for each of the 6 domains and provides a value ranging from 0 to 18. Higher scores indicate greater impairment. Positive change from baseline indicates greater impairment.
Time Frame: Baseline, Week 106
Population: Assessment was planned for Week 106 for this outcome measure, but no assessments were conducted at Week 106 due to early termination.
Arm/Group | Placebo | Aducanumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Global Statistical Test (GST) Composite Z-Score at Weeks 78 and 106
Description: GST z-score is an average of z-scores of CDR-SB, ADASCog13 and ADCS-ADL-MCI. CDR-SB assesses 3 cognitive (memory,orientation, judgment/problem-solving)and 3 functional(community affairs,home/hobbies,personal care) domains. Sum of Boxes method combines scores across 6 domains, ranging from 0-18(higher scores=greater impairment). ADAS-Cog13 evaluates cognitive tasks like word recall, naming, orientation and memory, with scores from 0-85 (higher scores=worse performance). ADCS-ADL-MCI rates 17 tasks (e.g.,shopping, preparing meal) and 1 basic task(dressing) with scores from 0-53 (higher scores=greater independence/healthy functioning). z-score>0 indicates greater impairment/worse performance for CDR-SB and ADASCog13 scales and improved functioning for ADCS-ADL-MCI. For ADCS-ADL-MCI, z-score were reversed (new reversed value=original value-1) to make interpretation consistent. The GST z-score of 0 indicates population mean and score>0 indicate greater impairment/worse performance.
Time Frame: Baseline, Weeks 78 and 106
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Placebo | Aducanumab
Number analyzed (Participants) | 3 | 4
z-score | 0.88 (0.116) | 0.48 (0.515)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to last follow-up visit (up to approximately 2 years 2 months)
Description: Safety analysis set included all randomized participants who had received at least 1 dose of study treatment (aducanumab or placebo). One participant in the placebo arm received drug. This participant was considered in Aducanumab group for safety analysis.
Arm/Group | Placebo | Aducanumab
All-Cause Mortality (participants affected / at risk) | 0/343 | 3/681
Serious Adverse Events (participants affected / at risk) | 23/343 | 59/681
Other Adverse Events (participants affected / at risk) | 127/343 | 359/681
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=343) | Aducanumab (N=681)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 0 | 2
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 0 | 7
Aphasia (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lacunar stroke (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 3
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2
Superficial siderosis of central nervous system (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 6
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Hypertensive emergency (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=343) | Aducanumab (N=681)
Covid-19 (Infections and infestations) | 19 | 49
Nasopharyngitis (Infections and infestations) | 26 | 42
Fall (Injury, poisoning and procedural complications) | 32 | 55
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 34 | 167
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 8 | 159
Dizziness (Nervous system disorders) | 17 | 42
Headache (Nervous system disorders) | 33 | 81
Superficial siderosis of central nervous system (Nervous system disorders) | 5 | 69

LIMITATIONS AND CAVEATS:
The study was terminated prematurely based on the sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally, the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor's Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of the Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT05310071/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT05310071/SAP_001.pdf